CLINICAL TRIAL: NCT01618019
Title: Effect of n-3 Polyunsaturated Fatty Acid Supplementation on Patients With Rheumatoid Arthritis
Brief Title: N-3 PUFA and Rheumatoid Arthritis in Korea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanyang University (Other)
Responsible Party: Principal Investigator, Yongsoon Park, Associate Professor, Hanyang University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: HYUH-C55; KRF-2010-000-8656 (Other Grant/Funding Number: KRF, Korean Government)
Record Dates: First submitted 2012-06-08; First posted 2012-06-13 (Estimated); Results first posted 2012-10-02 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-08

CONDITIONS: Rheumatoid Arthritis
Keywords: n-3 PUFA; rheumatoid arthritis; inflammation; eicosanoids; bone turnover markers
MeSH Terms: conditions — Arthritis, Rheumatoid; Inflammation | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- N-3 PUFA (Experimental): 5 capsules/day of n-3 PUFA, containing 2.09 g eicosapentaenoic acid and 1.165 g docosahexaenoic acid
  Interventions: Dietary Supplement: Omega-3 fatty acid
- Placebo (Placebo Comparator): 5 capsules/day of placebo containing sunflower with oleic acid (DSM Nutritional products, Switzerland)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Omega-3 fatty acid — 5 capsules/day of either n-3 PUFA, containing 2.09 g eicosapentaenoic acid and 1.165 g docosahexaenoic acid
  Other Names: Ropufa 75 n-3, DSM Nutritional products, Switzerland
  Arms: N-3 PUFA
Dietary Supplement: Placebo — 5 capsules/day of placebo containing sunflower with oleic acid (DSM Nutritional products, Switzerland)
  Arms: Placebo

SUMMARY:
The purpose of this study is to see if supplementation of n-3 polyunsaturated fatty acid (PUFA) can be beneficial for the patients with rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with rheumatoid arthritis diagnosed based on American College of Rheumatology guideline and receiving NSAID, glucocorticoids, or DMARD were eligible if the dosage had been stable for at least 3 months prior to entering the study.

Exclusion Criteria:

* Patients were excluded if they were pregnant, lactating, under the age of 18 or over age 80, taking supplements containing n-3 PUFA, white blood cell (WBC) ≤ 3.5 × 109/L, hemoglobin (Hb) ≤ 8.5 g/dL, platelet ≤ 100 × 109/L, creatinine ≥ 2.0 mg/dL, and aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥ 2.5 times upper limit of normal.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2010-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yongsoon Park, PhD, Principal Investigator — Hanyang University
Locations (1):
- Hanyang university hospital, Seoul, South Korea

REFERENCES:
- [Derived] Park Y, Lee A, Shim SC, Lee JH, Choe JY, Ahn H, Choi CB, Sung YK, Bae SC. Effect of n-3 polyunsaturated fatty acid supplementation in patients with rheumatoid arthritis: a 16-week randomized, double-blind, placebo-controlled, parallel-design multicenter study in Korea. J Nutr Biochem. 2013 Jul;24(7):1367-72. doi: 10.1016/j.jnutbio.2012.11.004. Epub 2013 Jan 17. PMID 23333088

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with rheumatoid arthritis diagnosed based on American College of Rheumatology guideline were recruited from Hanyang university hospital in Seoul, Eulji university hospital in Daejun, Catholic university hospital in Daegu, and Maryknoll medical center in Busan between Dec 2010 and Dec 2011.
Pre-assignment Details: Patients receiving NSAID, glucocorticoids, or DMARD were eligible if the dosage had been stable for at least 3 months prior to entering the study.
Period: Overall Study
Arm/Group | N-3 PUFA | Placebo
Started | 55 | 54
Completed | 41 | 40
Not Completed | 14 | 14
Not completed — Withdrawal by Subject | 14 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | N-3 PUFA | Placebo | Total
Number analyzed (Participants) | 55 | 54 | 109
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 51 | 52 | 103
  >=65 years | 4 | 2 | 6
Age Continuous [Mean (Standard Deviation); unit: years] | 49.51 (10.71) | 48.67 (8.91) | 49.09 (9.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 50 | 101
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 55 | 54 | 109

OUTCOME MEASURES:

1. Primary Outcome: Dose of NSAID
Description: Daily non-steroidal anti-inflammatory drug (NSAID) requirements as mg/day
Time Frame: 16 week
Population: Per-protocol analysis (except for drop out patients) Measurement of NSAID requirements at 16 weeks, except for 10 in N-3 PUFA and 6 in placebo.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | N-3 PUFA | Placebo
Number analyzed (Participants) | 41 | 40
mg | 319.72 (407.10) | 301.58 (337.18)

2. Secondary Outcome: Duration of Morning Stiffness
Description: Duration of morning stiffness means that patients with rheumatoid arthritis feel those joints stiff when they wake up in the morning.
Time Frame: 16 week
Population: Per-protocol analysis (except for drop out patients) Measurement of Morning stiffness assessment at 16 weeks, except for 16 in N-3 PUFA and 16 in placebo
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | N-3 PUFA | Placebo
Number analyzed (Participants) | 41 | 40
minutes | 40.10 (79.28) | 17.55 (29.20)

3. Secondary Outcome: Physician's Global Assessment
Description: Physician's global assessment is ranged from 0 to 10 by the assessing physician.
  (0= no pain; 10= very severe pain)
Time Frame: 16 week
Population: Per-protocol analysis (except for drop out patients) Measurement of Physician's global assessment at 16 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N-3 PUFA | Placebo
Number analyzed (Participants) | 41 | 40
units on a scale | 1.88 (1.83) | 1.60 (1.75)

4. Secondary Outcome: Patient's Global Assessment
Description: Patient's global assessment is patient self-assessed disability. (0= better condition; 10= very worse condition)
Time Frame: 16 week
Population: Per-protocol analysis (except for drop out patients) Measurement of Patient's global assessment at 16 week.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N-3 PUFA | Placebo
Number analyzed (Participants) | 41 | 40
units on a scale | 4.00 (2.57) | 4.01 (2.22)

5. Secondary Outcome: Pain Scale
Description: Pain scale is ranged from 0 to 100. (0= no pain; 100= severe pain)
Time Frame: 16 week
Population: Per-protocol analysis (except for drop out patients) Measurement of Pain scale at 16 week.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N-3 PUFA | Placebo
Number analyzed (Participants) | 41 | 40
units on a scale | 35.85 (26.41) | 28.75 (20.90)

6. Secondary Outcome: Osteocalcin Concentration
Description: serum Osteocalcin concentration as nmol/L
Time Frame: 16 week
Population: Per-protocol anlysis (except for drop out patients) serum Osteocalcain concentration at 16 week
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | N-3 PUFA | Placebo
Number analyzed (Participants) | 41 | 40
nmol/L | 0.90 (0.36) | 0.87 (0.29)

7. Secondary Outcome: BSAP Concentration
Description: serum bone specific alkaline phosphatase concentration as U/L
Time Frame: 16 week
Population: Per-protocol analysis (except for drop out patients) serum bone specific alkaline phosphatase concentration at 16 week
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | N-3 PUFA | Placebo
Number analyzed (Participants) | 41 | 40
U/L | 12.31 (4.85) | 12.27 (5.45)

8. Secondary Outcome: CTX Concentration
Description: serum C-terminal telopeptide of type 1 collagen concentration as nmol/L
Time Frame: 16 week
Population: Per-protocol analysis (except for drop out patients) serum C-terminal telopeptide of type 1 collagen concentration at 16 week
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | N-3 PUFA | Placebo
Number analyzed (Participants) | 41 | 40
nmol/L | 1.41 (1.05) | 1.35 (1.00)

ADVERSE EVENTS:
Arm/Group | N-3 PUFA | Placebo
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/54
Other Adverse Events (participants affected / at risk) | 0/55 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes